CLINICAL TRIAL: NCT00963339
Title: Age-Related Macular Degeneration (AMD) - Usability Study
Acronym: AMD
Status: Completed | Type: Observational
Sponsor: Notal Vision Ltd. (Industry)
Responsible Party: Osnat Ehrman/Clinical manager, Notal Vision
Organization: Notal Vision Inc. (Industry)
Other Study IDs: US02
Record Dates: First submitted 2009-08-20; First posted 2009-08-21 (Estimated); Last update posted 2010-09-23 (Estimated); Status verified 2010-09

CONDITIONS: Age Related Macular Degeneration
Keywords: AMD
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Dry AMD: subjects diagnosed as intermediate AMD in at least one eye
  Interventions: Device: Foresee Home

INTERVENTIONS:
Device: Foresee Home — Home Monitoring

SUMMARY:
The purpose of this study is to evaluate the usability of the Foresee Home device with intermediate AMD patients.

DETAILED DESCRIPTION:
The AMD usability study is a prospective, longitudinal, multi-center, observational study of patients diagnosed with intermediate (dry) AMD who have been asked by their doctor to use the ForeseeHomeTM device to record the natural progression of their AMD, including conversion from the dry to wet stage.

ELIGIBILITY:
Inclusion criteria

* Subjects diagnosed as intermediate AMD in at least one eye
* Visual Acuity (VA) with habitual correction <20/60 in the study eye
* Qualified in the clinic to use the device
* Ability to speak, read and understand instructions in English
* Subjects with ability to comprehend and sign the informed consent/authorization

Exclusion criteria

* Evidence of macular disease other than AMD or glaucoma in the study eye
* Presence of any significant media opacity that precludes a clear view of the macular area as identified in the study eye by biomicroscopy
* Any non-macular related ocular surgery performed within 3 months prior to study entry in the target eye

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Intermediate AMD
Sampling Method: Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2009-09; Primary Completion 2009-12 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Successful unpacking and installation | 3 months
Successful self tutorial performance | 3 months
Ability of the subjects to operate the device as define by a successful test completion | 3 months

SECONDARY OUTCOMES:
Evaluate the success rate of the interactive tutorial as defined by a reliable test result. | 3 month

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Roth, MD, Principal Investigator — Vitreos retina center - NJ